CLINICAL TRIAL: NCT01903655
Title: Study of the Telomere-telomerase System and the Expression of Candidate Genes in the Leukocytes of Patients With Depressive Disorder: Search for Peripheral Markers of Somatic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Chauvet PHRC IR 2009
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

ARMS (3):
- patients with a first episode of major depressive disorder (Other): a group of patients with a first episode of major depressive disorder according to DSM-IV-TR including depressive episodes with melancholic features
  Interventions: Other: telomere length
- patients with recurrent depressive disorder (Other): a group of patients with recurrent depressive disorder according to DSM-IV-TR including depressive episodes with melancholic features (at least three episodes of depression)
  Interventions: Other: telomere length
- control group (Other): patient with no depressive disorder during the study period and no psychiatric history
  Interventions: Other: telomere length

INTERVENTIONS:
Other: telomere length

SUMMARY:
The mechanisms of oxidative stress and inflammation involved in mood disorders are factors of chronicity and severity. These mechanisms induce a phenomenon of accelerated cellular senescence and are reflected by alterations in systemic gene expression detectable in leukocytes in peripheral blood. The genetic markers of these mechanisms are clinically significant markers. The identification of new genetic markers will make it possible to improve evaluations of the severity and somatic consequences of depressive syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have given their written informed consent
* absence of a diagnosis of major depressive disorder throughout the study and no history of psychiatric disorders
* diagnosis of a first episode of a major depressive disorder
* diagnosis of a recurrent major depressive disorder (at least three episodes) with or without resistance to therapy

Remarks:

* the diagnosis of major depressive disorder with characteristics of melancholy must be clearly mentioned in the case report form but is not a reason for not being included in the study
* the presence of a recent or older attempted suicide must lead to a careful clinical assessment of the diagnosis of depressive disorder and must be clearly mentioned in the case report form.

Exclusion Criteria:

* Persons not covered by the national Health Insurance Agency
* Psychotic or bipolar disorders
* Severe personality disorders
* cardiovascular disease, proven inflammatory disease and cancer
* persons unable to give their consent personally,
* persons in emergency situations,
* pregnant women,
* breast-feeding women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-04 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Telomere length | participants will be followed for the duration of hospital stay, an expected average of 6 months

SECONDARY OUTCOMES:
level of oxidative stress. | participants will be followed for the duration of hospital stay, an expected average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Result] Teyssier JR, Chauvet-Gelinier JC, Ragot S, Bonin B. Up-regulation of leucocytes genes implicated in telomere dysfunction and cellular senescence correlates with depression and anxiety severity scores. PLoS One. 2012;7(11):e49677. doi: 10.1371/journal.pone.0049677. Epub 2012 Nov 21. PMID 23185405